CLINICAL TRIAL: NCT03164681
Title: Red Blood Cell Distribution Width as a Predictor Marker of Contrast Induced Nephropathy in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Red Blood Cell Distribution Width as a Marker of Contrast Induced Nephropathy in Patients With Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherly Boshra, Principal Investigator, Assiut University
Other Study IDs: RDWCIN
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Contrast-induced Nephropathy
Keywords: sheerly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood ,serum,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contrast Induced Nephropathy is an acute renal insufficiency defined as a 25% or 0.5 mg/dl increase over the baseline of the serum creatinine level 24 h to 72 h after intravascular administration of a contrast agent.

DETAILED DESCRIPTION:
Contrast Induced Nephropathy has been introduced an important complication after coronary angiography and Percutaneous Coronary Intervention .

The development of Contrast Induced Nephropathy after Percutaneous Coronary Intervention is associated with poor clinical outcomes including prolonged hospitalization, increased costs, increased rates of end-stage renal failure, myocardial infarction, repeat revascularization, and short- and long-term mortality.

Contrast Induced Nephropathy follows decreased renal perfusion and administration of nephrotoxic medications as the third most common cause of renal insufficiency during hospitalization.

Patients with acute coronary syndrome have a 3-fold higher risk of developing Contrast Induced Nephropathy .Therefore ,predicting contrast nephropathy and initiating therapeutic preventive strategies are very important.

Red Blood Cell Distribution Width is a quantitive marker of the variability on size of erythrocyte.

It is a routine assay of Complete Blood Count that doesn't require an additional cost, that is calculated by dividing the standard deviation of the mean cell size by the Mean Corpuscular Volume of the red cells and multiplying by 100 to convert to a percentage.

Normal range of Red Blood Cell Distribution Width 11-16%. Increased Red Blood Cell Distribution Width means increased variability in red blood cell size owing to ineffective erythrocyte production, which is associated with indices of inflammation and pro-inflammatory cytokines such as interleukin-6 .

On the other hand, suggested mechanisms underlying Contrast Induced Nephropathy include cytotoxic effects, factors that affect renal hemodynamic, and regional hypoxia.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients who underwent percutaneous coronary intervention either elective or emergency.

Exclusion Criteria:

1. End stage renal disease with glomerular filtration rate less than 30 ml/1.73.
2. Patient known allergy to contrast agents.
3. Left ventricular ejection fraction below 30%.
4. Presence of infection
5. A recent history of contrast administration in the previous month.
6. Patient known to have thyroid disease.
7. History of malignancy.
8. Patient known to have Autoimmune disease.
9. Decompensated liver cirrhosis
10. Cardiogenic shock.
11. Anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Contrast Induced Nephropathy | 48 Hours
  Percentage of patients with raised serum creatinine 25% or 0.5 mg/dl over baseline serum creatinine within 48 hour after contrast administration

CONTACTS AND LOCATIONS:
Overall Officials: sherly boshra, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehran R, Nikolsky E. Contrast-induced nephropathy: definition, epidemiology, and patients at risk. Kidney Int Suppl. 2006 Apr;(100):S11-5. doi: 10.1038/sj.ki.5000368. PMID 16612394
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Background] Bartholomew BA, Harjai KJ, Dukkipati S, Boura JA, Yerkey MW, Glazier S, Grines CL, O'Neill WW. Impact of nephropathy after percutaneous coronary intervention and a method for risk stratification. Am J Cardiol. 2004 Jun 15;93(12):1515-9. doi: 10.1016/j.amjcard.2004.03.008. PMID 15194023
- [Background] Nash K, Hafeez A, Hou S. Hospital-acquired renal insufficiency. Am J Kidney Dis. 2002 May;39(5):930-6. doi: 10.1053/ajkd.2002.32766. PMID 11979336
- [Result] Tepel M, Aspelin P, Lameire N. Contrast-induced nephropathy: a clinical and evidence-based approach. Circulation. 2006 Apr 11;113(14):1799-806. doi: 10.1161/CIRCULATIONAHA.105.595090. No abstract available. PMID 16606801
- [Result] Seeliger E, Sendeski M, Rihal CS, Persson PB. Contrast-induced kidney injury: mechanisms, risk factors, and prevention. Eur Heart J. 2012 Aug;33(16):2007-15. doi: 10.1093/eurheartj/ehr494. Epub 2012 Jan 19. PMID 22267241